CLINICAL TRIAL: NCT05530109
Title: Study of Attentional Disorders in Patients Suffering From Idiopathic Generalized Epilepsy.
Acronym: ATTENTIONEPIG
Status: Terminated | Type: Observational
Why Stopped: IP's decision
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2021_0848; 2022-A00263-40 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2022-07-08; First posted 2022-09-07 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Idiopathic Generalized Epilepsy
Keywords: Attention; Epilepsy; Connectivity; EEG
MeSH Terms: conditions — Epilepsy, Idiopathic Generalized; Epilepsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with idiopathic generalised epilepsy
  Interventions: Other: Neuropsychological screening and high resolution EEG recording
- healthy controls: age- and sex-matched healthy controls
  Interventions: Other: Neuropsychological screening and high resolution EEG recording

INTERVENTIONS:
Other: Neuropsychological screening and high resolution EEG recording — Each participant will be assessed with a battery of neuropsychological tests including Epitrack, the Raven's progressive matrice, the MoCA, the D2-R test, the BDI-II test, the STAI and the Qolie-31. Then, a prolonged EEG recording at rest and during an attentional task (the ANT) will be realized

SUMMARY:
Attentional disorders have been reported in neuropsychological studies evaluating patients suffering from generalized idiopathic epilepsy, but the data are disparate (in terms of test protocol). We aim to describe attentional and executive function disorder in IGE thanks to the Epitrack scale, validated in this specific population. Our secondary objective is to study the dynamic of cortical activity during an attentional task (the ANT), in order to describe the alteration of cortical networks in epileptic patients presenting with attentional disturbance.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic generalized epilepsy followed-up during at least 2 years
* At least one antiepileptic drug medication
* No cognitive decline (MoCA score >26)
* Absence of concomitant pathology that could interfere with the purpose of the study.
* Be affiliated to the social security system
* Have signed an informed consent

Exclusion Criteria:

* Pregnancy
* Not able to give consent (Article 1121-8 of the CSP) Vulnerable person Being deprived of liberty by judicial or administrative decision (Article L 1121-6 of the CSP) Have a high probability of not respecting the protocol or of abandoning the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients from the clinical neurophysiology department of the Lille University Hospital, a reference centre for the follow-up of rare epilepsies.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2022-04-26 (Actual); Primary Completion 2025-04-25 (Actual); Study Completion 2025-04-25 (Actual)

PRIMARY OUTCOMES:
Epitrack scale score | At 1 month after inclusion
  EPITrack-Score shows the performance of attention and executive functions. Higher values indicate a better performance. scale from 9-49 (9 worst score - 49 best score)

SECONDARY OUTCOMES:
Raven's progressive matrice scores | At 1 month after inclusion
  cortical source connectivity patterns.
Montreal Cognitive Assessment (MoCA) score | At 1 month after inclusion
  Cognitive function was assessed by using MoCA score. Cognitive impairment was considered present when MoCA scores were <26 .
D2-R test score | At 1 month after inclusion
  cortical source connectivity patterns.
BDI-II score | At 1 month after inclusion
  Anxiety-depressive symptoms score Beck Depressive Inventory Questionnaire (BDI-II) (score), higher scores mean worse outcome, value minimum of 0 maximum 63
STAI scale | At 1 month after inclusion
  Anxiety-depressive symptoms score The State-Trait Anxiety Inventory (STAI) is a self-questionnaire, 20 questions, a score is calculated, ranging from 20 to 80, a high score indicating the presence of anxiety.
quality of life using the Qolie-31 self questionnaire | At 1 month after inclusion
  Quality Of Life In Epilepsy-Problems questionnaire (QOLIE31-P) questionnaire has been developed specifically to measure the quality of life of patients with epilepsy. The score ranges from 0 to 100 points. Higher scores reflect better quality of life; lower ones, worse quality of life.
High resolution Electro Encephalo Gram functional connectivity markers at rest and during the ANT task | At 1 month after inclusion
  limited number of reproducible resting activity patterns, brain networks involved in the absence of task performance

CONTACTS AND LOCATIONS:
Overall Officials: Philippe DERAMBURE, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hopital Roger Salengro, CHU Lille, Lille, France